CLINICAL TRIAL: NCT01421407
Title: Efficacy and Safety of High Intensity Focused Ultrasound (HIFU) Device to Treat Uncontrolled Secondary Hyperparathyroidism in Chronic Haemodialysis Patients
Brief Title: Efficacy and Safety of High Intensity Focused Ultrasound (HIFU) Device to Treat Secondary Hyperparathyroidism
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Theraclion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIFU/E/HPT2/Jan2011
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Secondary Hyperparathyroidism; End Stage Renal Disease; Parathyroid Hyperplasia
Keywords: Secondary hyperparathyroidism; End stage renal disease; Parathyroid hyperplasia; High Intensity Focused Ultrasound
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Intensity Focused Ultrasound (Active Comparator)
  Interventions: Device: Ultrasonic ablation device
- Control group (No Intervention)

INTERVENTIONS:
Device: Ultrasonic ablation device — High Intensity Focused Ultrasound treatment
  Other Names: TH-One
  Arms: High Intensity Focused Ultrasound

SUMMARY:
Secondary hyperparathyroidism (sHPT) is common in patients with chronic kidney disease (CKD), including those who are undergoing long-term haemodialysis treatment. sHPT is characterized by persistently elevated levels of parathyroid hormone (PTH) and major disturbances in phosphorus and calcium metabolism. When glomerular filtration rate (GFR) falls, the phosphorus clearance decreases significantly, leading to phosphorus retention. The resulting hyperphosphatemia is thought to be one of the principal causes of secondary hyperparathyroidism which is a very early complication of patients with CKD. Its diagnosis and treatment is crucial in the management of such patients.The treatment of the sHPT of CKD's patient includes dietary phosphate restriction, the use of phosphate binders, correction of hypocalcaemia, the use of vitamin D and its derivatives. The calcimimetic agent cinacalcet hydrochloride may be also used in combination with vitamin D. While the majority of patients can be controlled in this way, medical therapy is not always successful in achieving adequate control of secondary hyperparathyroidism. Oral medications (calcimimetics, recently developed phosphate binders, and active vitamin D derivatives amount to very high monthly costs, and have efficacy limitations as well as side-effects.

HIFU may become a valuable alternative treatment that help control secondary hyperparathyroidism in selected patients presenting with enlarged parathyroid gland(s) visible at ultrasonography,.

The aim of this study is to evaluate the efficacy and safety of HIFU treatment in chronic haemodialysis patients with secondary hyperparathyroidism presenting with enlarged parathyroid gland(s) which are visible at ultrasonography and for whom medical therapy has been unsuccessful.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years or older with end stage renal disease (ESRD) on thrice-weekly stable haemodialysis since at least 3 months with biochemically uncontrolled secondary hyperparathyroidism.
* PTH > 800 pg/ml with serum calcium > 8.4 mg/dl shown by three measurements obtained within a 30-day screening period, in spite of established maintenance dose for at least 3 months of Cinacalcet (>30mg/day) with or without vitamin D .
* Patients who underwent subtotal parathyroidectomy or total parathyroidectomy without autotransplantation and have recurrent secondary hyperparathyroidism, are eligible provided that they meet all the other inclusion criteria and exclusion criteria.
* Patients with one or two enlarged parathyroid glands, located with ultrasonography and with one or two over-active glands at sestamibi scintigraphy.

Exclusion Criteria:

* Primary or Tertiary Hyperparathyroidism (hyperparathyroidism after kidney transplantation).
* Serum total calcium (corrected for albumin) < 8.4 mg/dl (2.1 mmol/l)
* Serum ionized calcium < 1 mmo/l.
* Patient who underwent total parathyroidectomy with autotransplantation.
* Known history of parathyroid or other neoplasias in the neck region.
* History of neck irradiation
* Patients with abnormal vocal cord mobility revealed by indirect laryngoscopy
* Patients with enlarged parathyroid glands, not accessible to HIFU treatment.
* Head and/or neck disease that prevents hyperextension of neck. - Major surgery or arterio-venous fistula clotting in the last 3 months or major surgery projected in the subsequent 4 months.
* Pregnant or lactating woman.
* Patients whose concurrent illnesses, disability, or geographical residence would hamper attendance at required study visit.
* Patient receiving drugs such as flecainide, thioridazine, and most tricyclic antidepressants.
* Patients who are currently participating in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with a reduction from baseline of at least 30% in mean serum iPTH levels at 6 months after the last HIFU session and continuation of optimal medical therapy. | 6 months after the last HIFU session

SECONDARY OUTCOMES:
Proportion of patients with a serum PTH in the KDIGO in the recommended range (approximately two to nine times the upper normal limit for the assay) | at 6 months after last HIFU session

CONTACTS AND LOCATIONS:
Overall Officials: Angel Luis Martin DE FRANCISCO, Pr, Principal Investigator — Hospital Universitario Valdecilla. Santander. Spain
Locations (3):
- Italy (2):
  - Ospedale generale regionale "Miulli", Acquaviva delle Fonti
  - Ospedale Maggiore Policlinico Mangiagalli e Regina Elena, Milan
- Hospital Universitario Marquès de Valdecilla, Santander, Cantabria, Spain